CLINICAL TRIAL: NCT07129746
Title: Comparison Between Metallic Clip Ligation and Suture Ligation of Appendicular Stump in Laparoscopic Appendectomy, a Randomized Control Trial
Brief Title: Comparison Between Metallic Clip Ligation and Suture Ligation of Appendicular Stump in Laparoscopic Appendectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinnah Hospital (Other)
Responsible Party: Principal Investigator, MUHAMMAD SAUD IQBAL, Post-graduate resident, Principal Investigator, Jinnah Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: Jinnah Hospital Lahore
Record Dates: First submitted 2025-08-03; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Laparoscopic Appendectomy
Keywords: Appendicitis; Laparoscopy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Patients undergoing metallic clip ligation (Active Comparator): One of the standard methods of appendicular stump ligation
  Interventions: Device: Metallic clip ligation of the appendicular stump
- Group B - Patients undergoing suture material ligation of appendicular stump (Experimental): A feasible testing method with an anticipated increase in the length of surgery
  Interventions: Device: Suture ligation of appendicular stump

INTERVENTIONS:
Device: Metallic clip ligation of the appendicular stump — The group A patients will be having the appendicular stump ligated using the metallic clip, and assessed in terms of length of surgery and associated intra operative complications.
  Arms: Group A - Patients undergoing metallic clip ligation
Device: Suture ligation of appendicular stump — The appendicular stump in the second arm will be ligated using appropriate suture material and assessed in terms of length of surgery and rate of intraoperative complications.
  Arms: Group B - Patients undergoing suture material ligation of appendicular stump

SUMMARY:
Laparoscopic appendectomy is the standard procedure for acute appendicitis. Among the various steps of the procedure one of the rate limiting step is the ligation of the appendicular stump which can be done using suture material, metallic clips and hem o loks. This study compares the effect the using metallic clips versus suture material in the ligation of appendicular stump in terms of length of surgery and associated intra-operative complications. The patients included will be within the age group of 15-60 years, with BMI of 18-28kg/m2, and with acute appendicitis of upto grade 3. The data will be analyzed using SPSS a p value of <0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders, within the age bracket of 15 years - 60 years.
2. With a BMI within the range of 18 - 28 kg/m2.
3. With a diagnosis made by a consultant surgeon and the grade of appendicitis upto 3.

Exclusion Criteria:

1. Patients with long standing comorbidities including chronic liver disease, diabetes mellitus, chronic kidney disease and hemorrhagic disorders.
2. Patients taking anticoagulants, carrier of active cases of Hepatitis B, C and/or HIV.
3. Patients on immunosuppression therapy. Diameter of appendicular stump of more than 10mm, perforated appendix, laparoscopic appendectomy converted to open appendectomy pelvic appendicitis and sub-hepatic appendicitis.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Length of surgery | Intraoperative
  The length of surgery will be measured in terms of minutes from the start of the pneumoperitoneum insufflation till the evacuation of the pneumoperitoneum at the conclusion of the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinnah Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
The individual patient data will not be shared with other researchers on the basis of keeping confidentiality of the patients since this is a small center localized study. The matter was discussed with the ethical review board and the study was agreed upon under the aforementioned condition.

REFERENCES:
- [Background] Lee JS, Hong TH. Comparison of various methods of mesoappendix dissection in laparoscopic appendectomy. J Laparoendosc Adv Surg Tech A. 2014 Jan;24(1):28-31. doi: 10.1089/lap.2013.0374. Epub 2013 Nov 8. PMID 24206120
- [Background] Sohn M, Agha A, Bremer S, Lehmann KS, Bormann M, Hochrein A. Surgical management of acute appendicitis in adults: A review of current techniques. Int J Surg. 2017 Dec;48:232-239. doi: 10.1016/j.ijsu.2017.11.028. Epub 2017 Nov 16. PMID 29155250